CLINICAL TRIAL: NCT02114658
Title: A Multi-center, Single-arm, Open-label Phase II Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Sorafenib in Japanese Patients With Anaplastic Thyroid Carcinoma or Locally Advanced or Metastatic Medullary Thyroid Carcinoma
Brief Title: Sorafenib Phase II Study for Japanese Anaplastic or Medullary Thyroid Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17073
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Thyroid Carcinoma
Keywords: Anaplastic and medullary thyroid carcinoma; Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Sorafenib 400 mg bid continuous dose
  Interventions: Drug: Sorafenib (Nexavar,BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar,BAY43-9006) — Sorafenib 400 mg will be administered orally,twice daily in a 28 day cycle

SUMMARY:
The objectives of this study are to evaluate safety, efficacy and pharmacokinetics of sorafenib for the treatment of Japanese patients with anaplastic thyroid carcinoma (ATC) or locally advanced or metastatic medullary thyroid carcinoma (MTC).

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with ATC (Anaplastic thyroid carcinoma) or locally advanced or metastatic MTC (medullary thyroid carcinoma)
* Not a candidate for surgery or radiotherapy with curative intent
* Histologically or cytologically confirmed ATC or MTC
* Measurable or non-measurable disease (but clinically evaluable) according to RECIST 1.1.
* Age >= 18 years
* Adequate bone marrow, liver and renal function to be conducted within 14 days prior to treatment
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Histologic subtypes of thyroid cancer other than anaplastic or medullary carcinoma
* Prior anti-cancer treatment with tyrosine kinase inhibitors, monoclonal antibodies (licensed or investigational) that target VEGF or VEGF (vascular endothelial growth factor) receptors or other targeted agents
* Prior chemotherapy for thyroid cancer (only one regimen is allowed)
* Major surgery, open biopsy, or significant traumatic injury within 30 days prior to enrollment in the study.
* Subjects with tracheal, bronchial or esophageal infiltration with significant risk of bleeding but without having received local treatment prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2016-08-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events as a measure of safety and tolerability | 6 months
Change in red blood cell count | Baseline and 6 months
Change in white blood cell count | Baseline and 6 months
Change in alanine aminotransaminase level (ALT) | Baseline and 6 months
Change in aspartate aminotransferase level (AST) | Baseline and 6 months
Change in blood pressure | Baseline and 6 months

SECONDARY OUTCOMES:
Best overall response based on RECIST 1.1 criteria | Baseline and every 56 days up to progressive disease,an expected average of 8 months
Plasma concentration of sorafenib | Cycle 2 Day 1
Progression-free survival (PFS) | Baseline to progression or death by any reason
Overall survival (OS) | Baseline to death by any reason
Response rate (RR) | Baseline and every 56 days up to progressive disease
  RR based on RECIST 1.1 criteria
Disease control rate (DCR) | Baseline and every 56 days up to progressive disease
  DCR based on RECIST 1.1 criteria
Maximum reduction from baseline in the target lesion size | Baseline and every 56 days up to progressive disease
Maximum percentage change of calcitonin and Carcinoembryonic antigen (CEA) values from baseline | Baseline and every 56 days up to progressive disease
  MTC subjects only

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Japan (5):
  - Kobe, Hyōgo
  - Matsumoto, Nagano
  - Bunkyo-ku, Tokyo
  - Koto-ku, Tokyo
  - Osaka